CLINICAL TRIAL: NCT00002480
Title: Phase I Study of 3-Dimensional Conformal Radiotherapy in Patients With Locally Advanced (Stage T2c and T3) Adenocarcinoma of the Prostate
Brief Title: Radiation Therapy in Treating Patients With Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Purpose: Treatment
Other Study IDs: 91-022; CDR0000077099 (Registry Identifier: PDQ (Physician Data Query)); NCI-V91-0102
Record Dates: First submitted 1999-11-01; First posted 2004-03-11 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy

INTERVENTIONS:
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Radiation therapy may be an effective treatment for prostate cancer.

PURPOSE: Phase I trial to study the effectiveness of radiation therapy in treating patients who have stage II or stage III prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of radiotherapy using 3-dimensional (3D) conformal techniques in patients with stage II or III adenocarcinoma of the prostate. II. Determine the morbidity of high-dose 3D conformal therapy in these patients.

OUTLINE: This is a dose escalation study. Patients undergo 3-dimensional conformal radiotherapy 4-5 days a week for at least 8 weeks. Cohorts of 20-40 patients receive escalating doses of radiotherapy until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which no more than 10% of patients experience dose-limiting toxicity. Patients are followed at 3 months, every 6 months for 5 years, and then annually thereafter.

PROJECTED ACCRUAL: A minimum of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Locally advanced (T2c-T3) adenocarcinoma of the prostate including: Bulky tumors confined to prostate (stage II) Tumors extending beyond capsule (stage III) PSA no greater than 20 ng/mL No regional lymph node involvement (by CT scan or surgical sampling) No distant metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 60-100% Life expectancy: Not specified Hematopoietic: WBC greater than 4,000/mm3 Platelet count greater than 100,000/mm3 Hemoglobin greater than 11 g/dL Hepatic: Not specified Renal: Not specified Other: No major medical or psychiatric illness that would preclude study No metallic pelvic prosthesis

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior biologic therapy Chemotherapy: No prior chemotherapy Endocrine therapy: Prior hormonal therapy allowed Radiotherapy: No prior radiotherapy (including pelvic irradiation) Surgery: No prior radical surgery for carcinoma of the prostate

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1991-02; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Zelefsky, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Leibel SA, Heimann R, Kutcher GJ, Zelefsky MJ, Burman CM, Melian E, Orazem JP, Mohan R, LoSasso TJ, Lo YC, et al. Three-dimensional conformal radiation therapy in locally advanced carcinoma of the prostate: preliminary results of a phase I dose-escalation study. Int J Radiat Oncol Biol Phys. 1994 Jan 1;28(1):55-65. doi: 10.1016/0360-3016(94)90141-4. PMID 7505776
- [Result] Leibel SA, Zelefsky MJ, Kutcher GJ, Burman CM, Kelson S, Fuks Z. Three-dimensional conformal radiation therapy in localized carcinoma of the prostate: interim report of a phase 1 dose-escalation study. J Urol. 1994 Nov;152(5 Pt 2):1792-8. doi: 10.1016/s0022-5347(17)32387-x. PMID 7933238
- [Result] Leibel SA, Zelefsky MJ, Kutcher GJ, Burman CM, Mohan R, Mageras GS, Ling CC, Fuks Z. The biological basis and clinical application of three-dimensional conformal external beam radiation therapy in carcinoma of the prostate. Semin Oncol. 1994 Oct;21(5):580-97. No abstract available. PMID 7939749
- [Result] Zelefsky MJ, Leibel SA, Burman CM, Kutcher GJ, Harrison A, Happersett L, Fuks Z. Neoadjuvant hormonal therapy improves the therapeutic ratio in patients with bulky prostatic cancer treated with three-dimensional conformal radiation therapy. Int J Radiat Oncol Biol Phys. 1994 Jul 1;29(4):755-61. doi: 10.1016/0360-3016(94)90563-0. PMID 8040021
- [Result] Zelefsky MJ, Leibel SA, Kutcher GJ, Kelson S, Ling CC, Fuks Z. The feasibility of dose escalation with three-dimensional conformal radiotherapy in patients with prostatic carcinoma. Cancer J Sci Am. 1995 Jul-Aug;1(2):142-50. PMID 9166467